

# Non-Interventional Study (NIS) Protocol

| Document Number: | c35930967-01 |
|---|---|
| BI Study Number: | 0205-0547 |
| BI Investigational Product(s): | Spiriva Respimat |
| Title: | Exacerbation Risk and Health Care Resource use among patients with asthma using ICS+Tiotropium versus ICS/LABA |
| Brief lay title: | Exacerbation Risk in Asthma |
| Protocol version identifier: | 1.0 |
| Date of last version of protocol: | 5/12/2021 |
| PASS: | No |
| EU PAS register<br>number: | Study not registered |
| Active substance: | Tiotropium 1.25 mcq. |
| Medicinal product: | N/A |
| Product reference: | N/A |
| Procedure number: | N/A |
| Marketing authorisation holder(s): | N/A |
| Joint PASS: | N/A |
| Research question and objectives: | To conduct a comparative effective analysis of patients using Tiotropium in combination with Inhaled Corticosteroids (ICS) versus those that use LABA medication in combination with ICS. |
| Country(-ies) of study: | US |

# Non Interventional Study Protocol BI Study Number 0205-0547


c35930967-01

| Proprietary confidential information © | 2021 Boenringer Ingelneim International GmbH or one or more of its affiliated companies |
|---|---|
| Author: | |
| Marketing authorisation holder(s): | N/A |
| In case of PASS, add: MAH contact person: | N/A |
| In case of PASS, add: | N/A |
| In case of PASS, add: | N/A |
| Date: | 5/12/2021 |
| | Proprietary confidential information Soehringer Ingelheim Group of companies. All rights reserved. r in part - be passed on, reproduced, published or otherwise used without prior written permission |

c35930967-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 1. TABLE OF CONTENTS

| TITLE PAGE | 1 |
|-----------------------------------------|----|
| 1. TABLE OF CONTENTS | 3 |
| 2. LIST OF ABBREVIATIONS | 5 |
| 3. RESPONSIBLE PARTIES | 6 |
| 4. ABSTRACT | 7 |
| 5 . AMENDMENTS AND UPDATES | 11 |
| 6. MILESTONES | 11 |
| 7. RATIONALE AND BACKGROUND | 11 |
| 8. RESEARCH QUESTION AND OBJECTIVES | 13 |
| 9. RESEARCH METHODS | 13 |
| 9.1 STUDY DESIGN | 13 |
| 9.2 SETTING | 16 |
| 9.2.1 Study sites | 16 |
| 9.2.2 Study population | 16 |
| 9.2.3 Study visits | 16 |
| 9.2.4 Study discontinuation | 16 |
| 9.3 VARIABLES | 16 |
| 9.3.1 Exposures | 16 |
| 9.3.2 Endpoints | 17 |
| 9.3.2.1 Primary endpoints | 17 |
| 9.3.2.2 Secondary endpoints | 17 |
| 9.3.3 Covariates | 17 |
| 9.4 DATA SOURCES | 18 |
| 9.5 STUDY SIZE | 19 |
| 9.6 DATA MANAGEMENT | 19 |
| 9.7 DATA ANALYSIS | 19 |
| 9.7.1 Main analysis | 19 |
| 9.7.3 Safety Analysis | 20 |
| 9.8 QUALITY CONTROL | 20 |
| 9.9 LIMITATIONS OF THE RESEARCH METHODS | 20 |

# Non Interventional Study Protocol BI Study Number 0205-0547

c35930967-01

| Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies 9.10 OTHER ASPECTS | 20 |
|---|---|
| 9.10.1 Data quality assurance | 20 |
| 9.10.2 Study records | 20 |
| 9.10.2.1 Source documents | 21 |
| 9.10.2.2 Direct access to source data and documents | 21 |
| 9.10.3 Completion of study | 21 |
| 9.10.4 Protocol deviations | 21 |
| 9.10.5 Compensation available to the patient in the event of study related injury | 21 |
| 10.PROTECTION OF HUMAN SUBJECTS | 21 |
| 10.1 STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONS | SENT<br>21 |
| 10.2 STATEMENT OF CONFIDENTIALITY | 21 |
| 11.MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS | 21 |
| 12.PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS | 21 |
| 13.REFERENCES | 22 |
| 13.1 PUBLISHED REFERENCES | 22 |
| 13.2 UNPUBLISHED REFERENCES | 23 |
| ANNEX 1. LIST OF STAND-ALONE DOCUMENTS | 23 |
| ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS | 23 |
| ANNEX 3. ADDITIONAL INFORMATION | 23 |
| ANNEX 4. REVIEWERS AND APPROVAL SIGNATURES | 23 |

Non Interventional Study Protocol BI Study Number 0205-0547

c35930967-01


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 2. LIST OF ABBREVIATIONS

ADR, Adverse Drug Reaction

AE, Adverse Event

AESI, Adverse Event of Special interest

CA, Competent Authority

CCDS, Company Core Data Sheet

CI, Confidence Interval

CML, Local Clinical Monitor

CRA, Clinical Research Associate

CRF, Case Report Form

CTCAE, Common Terminology Criteria for Adverse Events

CTP, Clinical Trial Protocol

eCRF, Electronic Case Report Form

ENCePP, European Network of Centres for Pharmacoepidemiology and Pharmacovigilance

FDA, Food and Drug Administration

GCP, Good Clinical Practice

GEP, Good Epidemiological Practice

GPP, Good Pharmacoepidemiology Practice

GVP, Good Pharmacovigilance Practices

IB, Investigator's Brochure

IEC, Independent Ethics Committee

IRB, Institutional Review Board

MAH, Marketing Authorization Holder

MedDRA, Medical Dictionary for Regulatory Activities

NIS, Non-Interventional Study

PASS, Post-Authorization Safety Study

SAE, Serious Adverse Event Adapt and complete as appropriate

001-MCS-90-118\_RD-23 (2.0) / Saved on: 02 Jul 2020

Non Interventional Study Protocol BI Study Number 0205-0547 

c35930967-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 3. RESPONSIBLE PARTIES

| Institution | Investigators | _ |
|-------------|---------------|---|
| BI | | |

Non Interventional Study Protocol BI Study Number 0205-0547


c35930967-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 4. ABSTRACT

| Name of compa | any: | | |
|---|---|---|---|
| Boehringer Inge | lheim | | |
| Name of finishe | ed medicinal | | |
| product: | | | |
| Spiriva Respima | ıt | | |
| Name of active | ingredient: | | |
| Tiotropium | | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 12 May 2021 | 0205-0547 | 1.0 | 12 May 2021 |
| Title of study: | Exacerbation Risk an | nd Health Care Resource use | among patients with |
| | asthma using ICS+T | iotropium versus ICS/LABA | |
| | Date: 05/12 2021 | | |
| | Version Number:1 | | |
| Rationale and | | ty level, patients with uncont | |
| background: | 1 | ased use of systemic corticost | · |
| | | nes recommend increasing the | |
| | | nation with long-acting β2-ag | , |
| | 1 | such as with a long-acting n | _ |
| | | e receptor antagonists (LTRA | |
| | | s have found similar respons | |
| | | etween patients on ICS/Tiotro | • |
| | _ | ommonly used in the real wo | |
| | 1 * | v available in the US since 20 | • |
| | _ | evidence data complimenting | |
| | | e to ICS/LABA. It is important | |
| | | on with ICS using real world | data to support further |
| | treatment recommen | | |
| Research | | rative analysis of patients usi | |
| question and | | haled Corticosteroids (ICS) v | ersus those that use LABA |
| objectives: | medication in combi | | |
| Study design: | | ntional study based on existing | C |
| | | roups: 1. ICS+Tio and 2. ICS | |
| | | sures, including demographi | |
| | | level defined using Charlson | |
| | _ | bidities not included in the C | |
| | | ol level, and other listed mea | |
| | | 1) technique, we will develop | |
| | - | ICS+Tio and ICS/LABA gro | oups. |
| Population: | 1. ICS+Tio; and 2: Io | CS/LABA. | |

# Non Interventional Study Protocol BI Study Number 0205-0547

c35930967-01

| Proprietary confidential | l information © 2021 Boehringe | er Ingelheim International GmbH o | r one or more of its affiliated companies |
|---|---|---|---|
| Name of compa | ny: | | |
| Boehringer Ingel | heim | | |
| | d medicinal product: | 1 | |
| Spiriva Respimai | _ | | |
| Name of active i | | | |
| Tiotropium | ingi cuiciic. | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| | 1 | | |
| Protocol date: 12 May 2021 Variables: | PSM Gender Age group Region ICS dose leve Control levee Rescue med Comorbiditi ICS history ICS history Season of in Index year Baseline all-hospitalizati Baseline ovenumber of u Insurance ty Hypertensio Gastroesoph Allergic Rhi Obesity Sinusitis Obstructive Cardiovascu Diabetes Renal failure Arthritis Osteoporosis Depression Cancer (excl | ables are ICS+Tio use volCS. Tell clication use es included in the Char (yes/no) duration dex date cause resource use (pre ons, or ER visits, or out er asthma medications erall medication history nique medications) pe n tageal reflux disease enitis sleep apnea tlar disease es luding basal cell carcine eumonia diagnosis f dyspnea during baselin | Ison Comorbidity Index esence vs. absences of tpatient visits) (use vs. no use) (polypharmacy defined as |
| | and ICD 10 | KU6.Ux | |

### Non Interventional Study Protocol BI Study Number 0205-0547

Study size:


c35930967-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies Name of company: Boehringer Ingelheim Name of finished medicinal product: Spiriva Respimat Name of active ingredient: Tiotropium Protocol date: Study number: Version/Revision: Version/Revision date: 12 May 2021 0205-0547 12 May 2021 1.0 Variables: Diagnosis of alcohol dependence during baseline identified using ICD 9 303.xx, 305.0x and ICD 10 F10.xx Smoking dependence during baseline identified using ICD 9 305.1 and ICD 10 F17.xx Regression In addition to the key independent variable of interest (ICS+TIO vs. ICS/LABA group), we will include time varying medication exposure as a covariate in the regression. We will utilize medical and pharmacy claim records from Data sources: and pharmacy claims data. This database is comprised of adjudicated claims for more than 150 million commercially insured and Medicare lives in the US.

There are 25,291 patients with a prescription claim for tiotropium

monotherapy, will be applied to arrive at the final sample.

(1.25mcg, October 2015-May 2020) identified for analysis and 1,125,657 patients with ICS/LABA prescription claims (July 2014-May 2020). After excluding patients with COPD there are 17,882 patients in the Tio group and 921,804 patients in the ICS/LABA group. Further inclusion-exclusion criteria as well as restricting the Tio group to those with concurrent ICS

001-MCS-90-118\_RD-23 (2.0) / Saved on: 02 Jul 2020

### Non Interventional Study Protocol BI Study Number 0205-0547


c35930967-01

| Proprietary confidentia | l information © 2021 Boehrin | nger Ingelheim International GmbH or | one or more of its affiliated companies |
|---|---|---|---|
| Name of compa | ny: | | |
| Boehringer Inge | lheim | | |
| Name of finishe | d medicinal product | : | |
| Spiriva Respima | t | | |
| Name of active<br>Tiotropium | ingredient: | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 12 May 2021 | 0205-0547 | 1.0 | 12 May 2021 |

#### Data analysis

Sample attrition at each step of the inclusion-exclusion criteria will be provided. We will develop the breakdown of the distribution of demographic, comorbidity, and baseline measures prior to and after the PSM (unmatched and matched cohorts). Significance of differences will be tested at P<0.05 for the matched cohort. Additionally, we will consider the use of standardized mean differences as noted above, in which SMD < 0.1 indicates balance. The primary endpoint measure is time to first severe exacerbation and severe exacerbation will be defined as a hospitalization or an ER visit with a primary diagnosis of asthma. We will calculate the time in days to first exacerbation. We will conduct Cox proportional hazards modeling to estimate the risk of exacerbation and provide corresponding KM curves for the primary endpoint. Exposure to each of the study comparators (ICS+Tio and ICS/LABA) will be recorded using time-varying covariates for all primary and secondary endpoints. ICS+Tio vs. ICS/LABA will be the key independent variable and medication exposure will be a covariate included in the regression. Secondary endpoints will include time (in days) to first moderate-orsevere exacerbation defined as use of systemic corticosteroid or a hospitalization or ER visit with a primary diagnosis of asthma. Cox PH and KM curves will be conducted for this secondary end point as well. We will also calculate and compare the rate of exacerbation, proportion of patients with exacerbations after 6 months and one year among the subpopulation of patients having at least 6 months and a one year of followup, respectively. We will report rates in patient-years to account for variable follow-up time. We will also compare the mean monthly (to account for variable follow-up time) per patient HCRU (all-cause and asthma related hospitalizations, ER visits, and outpatient visits) during the follow-up period, between the two groups. Proportions of patients with and without rescue medication use will be compared between the two groups as well.

c35930967-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 5. AMENDMENTS AND UPDATES

None

#### 6. MILESTONES

| Study design and core group alignment | Week 1-2 |
|---|---|
| Data receipt, extraction, cleaning and evaluation for protocol development | Week 2 |
| Study protocol draft | Week 4 |
| Study protocol final | Week 6 |
| IET/NPCC approval | Week 8/9 |
| Descriptive statistics draft | Week 11-12 |
| Multivariate analysis draft | Week 12-14 |
| Final results (Excel) | Week 16-17 |
| Study narrative report | Week 17-18 |

#### 7. RATIONALE AND BACKGROUND

Asthma is associated with a significant burden on the healthcare system. More than half the population of asthma patients remains uncontrolled despite therapy, and uncontrolled asthma is associated with greater economic and health care burden (Braido et al. 2013; Peters et al. 2007). Stepwise treatment approach depending on control and severity levels has been the corner stone of asthma therapy. Regardless of severity level, patients with uncontrolled asthma are prone to exacerbations, increased use of systemic corticosteroids, rescue medications, deteriorating lung function (Chung et al. 2014), reduced quality of life, and increased health care resource use. In such cases, guidelines recommend increasing the dose of ICS product or use of ICS in combination with long-acting β2-agonists (LABA), and/or other add-on therapy such as with a long-acting muscarinic antagonist (LAMA), leukotriene receptor antagonists (LTRA), biologics or oral corticosteroids. Treatment strategies that rely on step treatment may not always be sufficient in controlling asthma.

Given the unmet needs, other therapeutic options should be considered in this population. In investigating Tiotropium (Handihaler and Respimat) for the treatment of asthma, 6 clinical trials (found similar responses in lung function and exacerbations when comparing ICS/Tiotropium to ICS/LABA. In a randomized controlled trial of moderate asthma patients, Kerstjens et al 2015 reported a lower rate of exacerbations among patients with ICS/Tiotropium when compared to ICS/Salmeterol (ICS/LABA) however formal comparisons could not be made since the ICS/salmeterol group was included to provide a standard add-on active comparator and was not part of the inferential analysis. Kerstjens et al study concluded that "Once-daily tiotropium as add-on treatment to medium-dose inhaled corticosteroids provided significant improvements in lung function and asthma control that were similar to those recorded for twice-daily salmeterol. In summary, RCTs have found

Non Interventional Study Protocol BI Study Number 0205-0547 

c35930967-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies similar responses in terms of lung function and exacerbations between patients on ICS/Tiotropium and ICS/LABA.

# NHLBI recommendations: Stepwise approach for management of asthma in patients ≥12 years



In 2020 NHLBI updated the Asthma guidelines recommending low dose ICS+LAMA as an alternative in Steps 3 and 4 noting that" the majority of LAMA studies use a comparative efficacy design and thus, their clinical impact is not well understood in real-world settings." The NHLBI response highlighted the need for RWE to close this data gap. This proposed real world evidence (RWE) study will fill a data gap of assessing exacerbation differences with ICS/Tiotropium. ICS/LABA is very commonly used in the real world since 2003, and Tiotropium was only available in the US since 2016, so it's important we generate real world evidence data complimenting the ICS/Tiotropium RCT data as an alternative to ICS/LABA using real world data to support further treatment recommendations.

Non Interventional Study Protocol BI Study Number 0205-0547


c35930967-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 8. RESEARCH QUESTION AND OBJECTIVES

To conduct a comparative analysis of patients using Tiotropium in combination with Inhaled Corticosteroids (ICS) versus those that use LABA medication in combination with ICS.

#### 9. RESEARCH METHODS

#### 9.1 STUDY DESIGN

- 1. Patients with least two asthma diagnosis (ICD 9 CM: 493.xx or ICD 10: J45-J45.999) will be included.
- 2. Patients will be required to be concurrently on ICS+Tiotropium (specifically Tiotropium Respimat® 1.25 mcg) or ICS/LABA.
- 3. Patients with least two diagnosis of COPD at any time during the study period will be excluded.
- 4. Patients less than 12 years of age will be excluded.
- 5. Patients will be required to have enrollment for at least 6 months prior to ICS+Tio or ICS/LABA use.
- 6. Patients on biologics within 6 months prior to ICS+Tio or ICS/LABA use will be excluded.
- 7. Patients with prior Tio or ICS/LABA use during the 6-month baseline period will be excluded.
- 8. Patients with urinary bladder obstruction, urinary retention, and glaucoma will be excluded.
- 9. After the PSM process, unmatched patients will be excluded.

Patients will be classified into two groups based on the exposure on the index date: 1. ICS+Tio; and 2: ICS/LABA. The date of concurrent medication initiation will be defined as the index date based on the date of the first prescription claim defining their add-on medication. We will record various baseline measures, including demographics such as gender, age, and region, comorbidity level defined using Charlson Comorbidity Index (CCI), other specific comorbidities not included in the CCI (Table 1), inhaled medication use, and control level as defined in Table 1. Additionally, we will classify patients based on their daily ICS dose levels as 'low dose ICS', 'medium dose ICS', and 'high dose ICS'. The dose levels will be assigned per GINA 2020 criteria (Global Initiative for Asthma. Global Strategy for Asthma Management and Prevention 2020). Medications that are available with only two dose level indications will be tagged as 'low' for the lower of the two dose levels, and 'high' for the highest dose level.

### **Non Interventional Study Protocol** BI Study Number 0205-0547


c35930967-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies **Table 1: Baseline Parameters and Variable Definitions** 

| Variable Name and Type | Description and Definition | Covariate Adjustment Method |
|---|---|---|
| Demographics | Age (5-year increments), Gender, | PSM |
| Region | Region (Northeast, Midwest, South, West) | PSM |
| CCI | Charlson Comorbidity Index score | PSM |
| Inhaled medication use | Identified using unique claims during the baseline period | PSM |
| Control Status:<br>Not Well Controlled or<br>Well Control | "Not Well Controlled" if patient has any one of the following events • Prescription for OCS • Asthma-related ER • Asthma-related hospitalizations "Well controlled" if patient has none of the above events (Ref: Stempel JACI 2005) | PSM |
| ICS history | Defined by use of ICS monotherapy prior to index date | PSM |
| ICS history duration | Days on ICS monotherapy prior to index date | PSM |
| ICS dose level | Daily dose of ICS classified as low dose ICS,<br>medium dose ICS, and high dose ICS | PSM |
| Season | Season of cohort entry (Summer, Spring, Fall, Winter) | PSM |
| Index year | Year of the index date | PSM |
| All-cause resource use | All-cause hospitalizations, ER visits, outpatient visits | PSM |
| Other asthma medications | Leukotriene modifiers | PSM |
| Medication history | Polypharmacy calculated based on number of unique medications | PSM |
| Insurance type | Identified using payer type data field | PSM |
| Hypertension | Identified using appropriate ICD codes. Coded as binary (yes/no) variables | PSM |
| Allergic rhinitis | Identified using appropriate ICD codes. Coded as binary (yes/no) variables | PSM |
| Sinusitis | Identified using appropriate ICD codes. Coded as binary (yes/no) variables | PSM |
| Obstructive sleep apnea | Identified using appropriate ICD codes. Coded as binary (yes/no) variables | PSM |
| Gastro-esophageal reflux disease | Identified using appropriate ICD codes. Coded as binary (yes/no) variables | PSM |
| Obesity | Identified using appropriate ICD codes. Coded as binary (yes/no) variables | PSM |
| Cardiovascular disease | Identified using appropriate ICD codes. Coded as binary (yes/no) variables | PSM |
| Diabetes | Identified using appropriate ICD codes. Coded as binary (yes/no) variables | PSM |

### Non Interventional Study Protocol BI Study Number 0205-0547


c35930967-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Variable Name and Type | Description and Definition | Covariate Adjustment Method |
|---|---|---|
| Renal failure | Identified using appropriate ICD codes. Coded as binary (yes/no) variables | PSM |
| Arthritis | Identified using appropriate ICD codes. Coded as binary (yes/no) variables | PSM |
| Depression | Identified using appropriate ICD codes. Coded as binary (yes/no) variables | PSM |
| Osteoporosis | Identified using appropriate ICD codes. Coded as binary (yes/no) variables | PSM |
| Cancer (excluding basal cell carcinoma) | Identified using appropriate ICD codes. Coded as binary (yes/no) variables | PSM |
| Pneumonia | Identified using appropriate ICD codes. Coded as binary (yes/no) variables | PSM |
| Acute bronchitis | Identified using appropriate ICD codes. Coded as binary (yes/no) variables | PSM |
| Dyspnea | Identified using appropriate ICD codes. Coded as binary (yes/no) variables | PSM |
| Alcohol dependence | Identified using appropriate ICD codes. Coded as binary (yes/no) variables | PSM |
| Smoking dependence | Identified using appropriate ICD codes. Coded as binary (yes/no) variables | PSM |

Using propensity score matching (PSM) technique, we will develop matched cohorts of patients between the ICS+Tio and ICS/LABA groups. We will conduct 1:2 matching using nearest neighbor matching approach. Upon completion of matching, we will assess whether the cohorts are balanced by examining the statistically significant differences at p<0.05. We will also assess balance by calculating standardized mean differences (SMD). An SMD < 0.1 will be considered balanced. Follow-up time will be calculated between index date and 'Censor date' which will be defined as the date of either one of the following events: 1. Date of first exacerbation, 2. Date of medication switch, 3. Discontinuation of medication (defined as date of prescription claim plus days' supply, plus 50% additional days), 4. Enrollment end date, or 5. Last date available in the dataset/End of study period. In this "new user", study design, primary analysis will be an "as-treated" analysis. In order to attribute events and outcomes to patients during the time that they are exposed to treatment (based on dayssupply of prescription claims + a buffer window) as well as account for differences in intergroup adherence levels, we will use a time-varying covariate approach to classify drug exposure time for each comparator drug during follow up. This approach has been chosen to minimize bias based on potentially large differences in medication adherence rates, by only attributing outcomes to the time in which patients have medication in their possession based on days' supply as described below. For each individual study drug, we will identify and define medication exposure and non-exposure windows during the follow-up time for each medication using the date of prescription filled plus the days' supply listed on the prescription claim plus 50% additional days (to account for residual doses in canister, poor real-world adherence and latency of drug effects). For example, exposure start and stop dates

c35930967-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies for a patient with a prescription claim with 30 days supply on January  $1^{st}$  will be January  $1^{st}$  and February  $15^{th}$  respectively (30 days' supply +15 days). We will run sensitivity analyses on the exposure window using 0% and 100% additional days. These time varying exposure covariates will be included in the Cox PH regression.

If statistical differences are found after PSM, then the study team will make a determination to either include them as covariates in the regression analysis (Cox PH), or develop interaction terms to match on, or discontinue the study. In the event of study discontinuation, partial results (all analysis leading up to and including PSM) will be provided in a final report.

#### 9.2 SETTING

Please see section 9.1.

9.2.1 Study sites
Please see section 9.1 and 9.4

9.2.2 Study population Please see section 9.1.

9.2.3 Study visits *Not applicable* 

9.2.4 Study discontinuation

Boehringer Ingelheim reserves the right to discontinue the study overall or at a particular study site at any time for the following reasons:

- 1. Failure to meet expected enrolment goals overall or at a particular study site
- 2. Violation of Good Pharmacoepidemiology Practice (GPP), the study protocol, or the contract by a study site, investigator, or research collaborator, disturbing the appropriate conduct of the study

The investigator/the study site/research collaborator will be reimbursed for reasonable expenses incurred in case of study/site termination (except in case of the third reason).

#### 9.3 VARIABLES

#### 9.3.1 Exposures

The exposure variables are Tio use vs. LABA use in combination with ICS. The operational definitions are provided in the sections above. After PSM, the cohort group will be the key predictor for the Cox PH regression to assess the primary outcome.

c35930967-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.3.2 Endpoints

#### 9.3.2.1 Primary endpoints

The primary endpoint measure is time to first severe exacerbation. Severe exacerbations will be defined as:

- A hospitalization with a primary diagnosis of asthma or
- An ER visit with a primary diagnosis of asthma

#### 9.3.2.2 Secondary endpoints

Secondary endpoints will include:

- Time to first moderate-or-severe exacerbation
  - o Any systemic corticosteroid use or
  - o A hospitalization with a primary diagnosis of asthma or An ER visit with a primary diagnosis of asthma
- Proportion of patients with exacerbation
- Rate of exacerbation at 6 months and one year
- Proportions of patients with Health care resource utilization (HCRU). HCRU is defined as hospitalizations, emergency room (ER) visits, and outpatient visits during follow-up, all-cause and asthma related.
- Mean monthly HCRU (including frequency of hospitalizations, ER visits, OP visits)
- Proportion of patients with use of rescue medications (defined as patients with one or more SABA claims during the follow-up period)



#### 9.3.3 Covariates

The covariates included in the PSM will be

- Gender
- Age group
- Region
- ICS dose level
- Control level
- Rescue medication use
- Comorbidities included in the Charlson Comorbidity Index
- ICS history (yes/no)
- ICS history duration
- Season of index date
- Index year
- Baseline all-cause resource use (presence vs. absences of hospitalizations, or ER visits, or outpatient visits)
- Baseline other asthma medications (use vs. no use)

### Non Interventional Study Protocol BI Study Number 0205-0547


c35930967-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Baseline overall medication history (polypharmacy defined as number of unique medications)
- Insurance type
- Hypertension
- Gastroesophageal reflux disease
- Allergic Rhinitis
- Obesity
- Sinusitis
- Obstructive sleep apnea
- Cardiovascular disease
- Diabetes
- Renal failure
- Arthritis
- Osteoporosis
- Depression
- Cancer (excluding basal cell carcinoma)
- Baseline pneumonia diagnosis
- Baseline acute bronchitis diagnosis
- Diagnosis of dyspnea during baseline identified using ICD 9 786.0x and ICD 10 R06.0x
- Diagnosis of alcohol dependence during baseline identified using ICD 9 303.xx, 305.0x and ICD 10 F10.xx
- Smoking dependence during baseline identified using ICD 9 305.1 and ICD 10 F17.xx

In addition to the key independent variable of interest (ICS+TIO vs ICS/LABA group), we will include time varying medication exposure as a covariate in the regression.

#### 9.4 DATA SOURCES

We will utilize medical and pharmacy claim records from medical and pharmacy claims data. This database is comprised of adjudicated claims for more than 150 million commercially insured and Medicare lives in the US. Data between 2014 and 2020 will be extracted, with the first patient follow-up period for tiotropium 1.25 mcg dose patients starting in October of 2015. This longitudinal database allows documentation and analysis of the patient journey from diagnosis to intervention and follow-up. The database includes patients in the majority of three-digit zip codes and in every metropolitan statistical area of the US. It also covers data from 90% of US hospitals, 80% of all US doctors, and represents 85% of the Fortune 100 companies, with current HIPAA (Health Insurance Portability and Accountability Act) regulations. The database is constructed from a variety of geographic regions and employer groups and maintains a level of diversity while representing the overall trend in commercial health plan coverage. The underrepresentation of the population aged 65 years and older may affect external validity in the case of Medicare, Medicare Advantage or Medicaid patients.

Non Interventional Study Protocol BI Study Number 0205-0547 

c35930967-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

9.5 STUDY SIZE

There are 25,291 patients with a prescription claim for tiotropium (1.25mcg, October 2015–May 2020) identified for analysis and 1,125,657 patients with ICS/LABA prescription claims (July 2014-May 2020). After excluding patients with COPD there are 17,882 patients in the Tio group and 921,804 patients in the ICS/LABA group. Further inclusion-exclusion criteria as well as restricting the Tio group to those with concurrent ICS monotherapy, will be applied to arrive at the final sample.

#### 9.6 DATA MANAGEMENT

The data management plan is summarized below. Full details of the data management plan are documented in a separate NIS-Data Management and Review Plan (NIS-DMRP).

All established security and confidentiality procedures will be observed by BI and/or personnel who are assigned appropriate access to the data. Enrolment data, medical claims, and prescription claims will be accessed from the administrative claims dataset. The analyses will be performed on limited data sets that are void of member protected health information and all results were shared in aggregate form only.

#### 9.7 DATA ANALYSIS

#### 9.7.1 Main analysis

Sample attrition at each step of the inclusion-exclusion criteria will be provided. We will develop the breakdown of the distribution of demographic, comorbidity, and baseline measures prior to and after the PSM (unmatched and matched cohorts). Significance of differences will be tested at P<0.05 for the matched cohort. Additionally, we will consider the use of standardized mean differences as noted above, in which SMD <0.1 indicates balance of baseline covariates. The primary endpoint measure is time to first severe exacerbation and severe exacerbation will be defined as a hospitalization or an ER visit with a primary diagnosis of asthma. We will calculate the time in days to first exacerbation. Also, as part of the primary end point analysis, we will develop KM curves based on initial exposure and conduct time varying Cox proportional hazards modeling accounting for changes in exposure status over the follow up time to estimate the risk of exacerbation between ICS+Tio vs. ICS/LABA. Secondary endpoints will include a number of measures. We will calculate the time in days to first moderate-or-severe exacerbation defined as use of systemic corticosteroid or a hospitalization or ER visit with a primary diagnosis of asthma. KM curves based on initial exposure and time varying Cox PH models will be conducted for this secondary end point as well. We will also calculate and compare the rate of exacerbation, proportion of patients with exacerbations after 6 months and one year among the subpopulation of patients having at least 6 months and a year of follow-up, respectively. We will report rates in patient-years to account for variable follow-up time. We will also compare the mean monthly (to account for variable follow-up time) per patient HCRU (all-cause and asthma related hospitalizations, ER visits, and outpatient visits) during the follow-up period, between the two groups. Proportions of patients with and without rescue medication use will be compared between the two groups as well.

Non Interventional Study Protocol BI Study Number 0205-0547

c35930967-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



9.7.3 Safety Analysis

No Adverse Events are anticipated to be identified in this study.

#### 9.8 QUALITY CONTROL

The quality control, review, and monitoring plan are summarized below. Greater details are documented in the NIS-DMRP.

All programming will be quality controlled by two-step code checking by results generated will be reviewed internally by two co-investigators separately prior to finalization.

#### 9.9 LIMITATIONS OF THE RESEARCH METHODS

As with all studies utilizing claims data, there are certain limitations. The presence of a claim for a filled prescription or prescription absent claim does not indicate that the medication was consumed or that it was taken as prescribed. Medications filled over-the-counter or provided as samples by the physician will not be observed in the claims data. Patients with commercial health insurance may be different from those with non-commercial or without (commercial) health insurance, and hence study results may not be generalizable to the overall population. Population aged 65 years and older might be underrepresented, which may affect external validity in the case of Medicare, Medicare Advantage or Medicaid patients. Socioeconomic data is not available and can affect asthma outcomes. Since unmatched patients will be excluded, the results may not be generalizable to all patients. Some study measures and outcomes will include missing data and hence reduce the sample size. Patient misclassification, missing data, objective and reliable measurement of patient outcomes, and lack of detailed information regarding subjects' clinical history or clinical status during the study timeframe may undermine the accuracy of our study results.

#### 9.10 OTHER ASPECTS

None

9.10.1 Data quality assurance

A quality assurance audit/inspection of this study may be conducted by the sponsor or sponsor's designees or by Institutional Review Board (IRBs) / Independent Ethics Committee (IECs) or by regulatory authorities. The quality assurance auditor will have access to all medical records, the investigator's study-related files and correspondence, and the informed consent documentation of this study.

9.10.2 Study records NA

### Non Interventional Study Protocol BI Study Number 0205-0547


c35930967-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies 9.10.2.1 Source documents

NA

9.10.2.2 Direct access to source data and documents

NA

9.10.3 Completion of study

NA

9.10.4 Protocol deviations

NA

9.10.5 Compensation available to the patient in the event of study related injury

NA

#### 10.PROTECTION OF HUMAN SUBJECTS

Ethical approval is not required for this study.

# 10.1 STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT

NA

#### 10.2 STATEMENT OF CONFIDENTIALITY

NA

# 11.MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

Not applicable based on secondary use of data without any potential that any employee of BI or agent working on behalf of BI will access individually identifiable patient data.

# 12.PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

The rights of the investigator and of the sponsor with regard to publication of the results of this study are described in the investigator contract. As a general rule, no study results should be published prior to finalization of the Study Report.

Non Interventional Study Protocol BI Study Number 0205-0547

c35930967-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 13.REFERENCES

#### 13.1 PUBLISHED REFERENCES

P10-10772 Peters SP, Kunselman SJ, Icitovic N et al. Tiotropium bromide step-up therapy for adults with uncontrolled asthma.N. Engl. J. Med., 363 (2010), pp. 1715-1726

P11-09529 Bateman ED, Kornmann O, Schmidt P et al. Tiotropium is noninferior to salmeterol in maintaining improved lung function in B16-Arg/Arg patients with asthma J. Allergy Clin. Immunol., 128 (2011), pp. 315-322

P14-03600 Chung KF et al. International ERS/ATS Guidelines on definition evaluation and treatment of severe asthma. Eur Respir J 43, 343-373 (2014)

P15-01655 Kerstjens HA et al. Tiotropium or salmeterol as add-on therapy to inhaled corticosteroids for patients with moderate symptomatic asthma: two replicate, double-blind, placebo-controlled, parallel-group, active-comparator, randomised trials. Lancet Respiratory Medicine. 2015 May;3(5):367-76.

P15-10269 Feehan M et al. Adherence to controller asthma medications: 6-month prevalence across a US community pharmacy chain. Journal of Clinical Pharmacy and Therapeutics, 2015

P15-11415 Wechsler M, Yawn B, Fuhlbrigge A et al. Anticholinergic vs Long-Acting  $\beta$ -Agonist in Combination With Inhaled Corticosteroids in Black Adults With Asthma: The BELT Randomized Clinical Trial. JAMA. 2015 Oct 27;314(16):1720-30.

P18-01651 Zhang L, Huang G, Jin L et al. Therapeutic effects of a long-acting cholinergic receptor blocker, tiotropium bromide, on asthma.Med. Sci. Mon. Int. Med. J. Exp. Clin. Res., 24 (2018), pp. 944-950

P18-08471 Buhl R, FitzGerald JM, Busse W. Tiotropium add-on to inhaled corticosteroids versus addition of long-acting  $\beta$ 2-agonists for adults with asthma. Respiratory Medicine. 2018. 143. Pages 82-90.

P19-00715 Braido F. Failure in Asthma control: Reasons and Conseuqences. Scientifica 2013. 549252 (2013)

P20-04444 Chipps B, Mosnaim G, Mathur SK, et al. Add-on tiotropium versus step-up inhaled corticosteroid plus long-acting beta-2-agonist in real-world patients with asthma. Allergy Asthma Proc. 2020;41(4):248-255. doi:10.2500/aap.2020.41.200036

P20-10184 Global Initiative for Asthma. Global Strategy for Asthma Management and Prevention (online appendix, updated 2020)

https://ginasthma.org/wp-content/uploads/2020/04/GINA-2020-Appendix\_final-wms.pd f (access date: 6 November 2020); 2020

#### Non Interventional Study Protocol BI Study Number 0205-0547

c35930967-01


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies R16-0701 Peters SP, Jones CA, Haselkorn T, Mink DR, Valacer DJ, Weiss ST. Real- world Evaluation of Asthma Control and Treatment (REACT): findings from a national web-based survey. J Allergy Clin Immunol 119 (6) 1454-1461 (2007)

R21-2127 Wu A et al. Primary Adherence to Controller Medications for Asthma Is Poor. Ann Am Thorac Soc. 2015 Feb;12(2):161-6

R21-2128 Stempel, David A. et al. Patterns of asthma control: A 3-year analysis of patient claims

Journal of Allergy and Clinical Immunology, Volume 115, Issue 5, 935-939

### 13.2 UNPUBLISHED REFERENCES

NA

#### ANNEX 1. LIST OF STAND-ALONE DOCUMENTS

*Not applicable* 

#### ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS

*Not applicable* 

#### **ANNEX 3. ADDITIONAL INFORMATION**

None

#### ANNEX 4. REVIEWERS AND APPROVAL SIGNATURES

Signatures will be provided electronically via approval workflow in the DMS for submission documents.